CLINICAL TRIAL: NCT05436912
Title: Open-label, Nonrandomized, Single-dose, Parallel-group, Safety, Tolerance, and Pharmacokinetic Study of LOXO-292 Administered to Fasted Hepatically Impaired Male and Female Subjects and Fasted Matched-control Healthy Subjects
Brief Title: A Study of Effects of Selpercatinib in Hepatically Impaired Participants and Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17483; J2G-OX-JZJD (Other: Eli Lilly and Company); LOXO-RET-18022 (Other: Loxo Oncology, Inc.)
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Hepatic Impairment
MeSH Terms: interventions — selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 160 milligram (mg) Selpercatinib: Normal Hepatic Function (Experimental): 160 mg selpercatinib administered orally to healthy participants after at least a 2-hour fast on Day 1.
  Interventions: Drug: Selpercatinib
- 160 mg Selpercatinib: Mild Hepatic Impairment (Experimental): 160 mg selpercatinib administered orally to participants with mild hepatic impairment per Child-Pugh [CP] classification (CP Class A, score of 5 or 6) after at least a 2-hour fast on Day 1.
  Interventions: Drug: Selpercatinib
- 160 mg Selpercatinib: Moderate Hepatic Impairment (Experimental): 160 mg selpercatinib administered orally to participants with moderate hepatic impairment per CP classification (CP Class B, score of 7 to 9) after at least a 2-hour fast on Day 1.
  Interventions: Drug: Selpercatinib
- 160 mg Selpercatinib: Severe Hepatic Impairment (Experimental): 160 mg Selpercatinib administered orally to participants with severe hepatic impairment per CP classification (CP Class C, score of 10 to 15) after at least a 2-hour fast on Day 1.
  Interventions: Drug: Selpercatinib

INTERVENTIONS:
Drug: Selpercatinib — Administered orally.
  Other Names: LY3527723; LOXO-292

SUMMARY:
The main purpose of this study is to assess how selpercatinib gets into the blood stream and how long it takes the body to remove it when administered to participants with impaired hepatic function compared to healthy participants. Information about safety and tolerability will be collected. The study will last up to about 7 weeks, inclusive of screening period.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of non-childbearing potential who are agreeable to take birth control measures until study completion
* Males who are capable of fathering a child must agree to use one of the following methods of contraception from the time of the dose administration through 6 months after dose administration:

  * Male sterilization, with documented confirmation of surgical success. Male subjects will be surgically sterile for at least 90 days prior to Check-in (Day -1). If documentation is not available, male subjects must follow one of the contraception methods below:
  * Male condom with spermicide, or
  * For a female partner of male study participant:
  * Intrauterine device (IUD) (hormonal IUD; eg, Mirena®). Copper IUDs are acceptable (eg, ParaGard®);
  * Established use of oral, implanted, transdermal, or hormonal method of contraception associated with inhibition of ovulation; or
  * Bilateral tubal ligation.
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilograms per meter squared (kg/m²) and had a minimum weight of at least 50 kg at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), and blood and urine laboratory test results that are acceptable for the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Had blood loss of more than 500 milliliters (mL) within the previous 30 days of study screening
* Require treatment with inducers or inhibitors of cytochrome P450 (CYP) CYP3A within 14 days before the first dose of study drug through the end of treatment or early termination

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (7):
  - Orange County Research Institute, Anaheim, California
  - National Institute of Clinical Research, Monterey Park, California
  - Orange County Research Center, Tustin, California
  - Riverside Clinical Research, Edgewater, Florida
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - The Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 160 Milligram (mg) Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment
Started | 12 | 8 | 8 | 8
Received at Least One Dose of Study Drug | 12 | 8 | 8 | 8
Completed | 12 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 160 mg Selpercatinib: Normal Hepatic Function: 160 mg selpercatinib administered orally to healthy participants after at least a 2-hour fast on Day 1.
- 160 mg Selpercatinib: Mild Hepatic Impairment: 160 mg selpercatinib administered orally to participants with mild hepatic impairment per CP classification (CP Class A, score of 5 or 6) after at least a 2-hour fast on Day 1.
- Total: Total of all reporting groups
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment | Total
Number analyzed (Participants) | 12 | 8 | 8 | 8 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (5.6) | 59 (4.5) | 57 (9.0) | 53 (4.7) | 56 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 6 | 6 | 22
  Male | 6 | 4 | 2 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 1 | 3 | 6 | 19
  Not Hispanic or Latino | 3 | 7 | 5 | 2 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 1 | 4
  White | 11 | 6 | 8 | 7 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 8 | 8 | 36

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Selpercatinib
Description: PK: Cmax of selpercatinib was reported.
Time Frame: Predose (within 30 minutes), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, and 240 hours postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
nanogram per milliliter (ng/mL) | 898 (129.8) | 1170 (78.0) | 732 (185.6) | 952 (72.3)
Statistical Analysis 1: Comparison: 160 mg Selpercatinib: Normal Hepatic Function vs 160 mg Selpercatinib: Mild Hepatic Impairment; Test type: Other; p = 0.3601, t-test, 2 sided; Geometric Mean Ratio = 168.9, 90% CI 2-sided [61.3 to 465.3] — Geometric mean ratio for natural log transformed parameter (expressed as a percent) and 90% confidence interval for geometric mean ratio of natural log transformed parameter (expressed as a percent), natural log transformed back to the linear scale
Statistical Analysis 2: Comparison: 160 mg Selpercatinib: Normal Hepatic Function vs 160 mg Selpercatinib: Moderate Hepatic Impairment; Test type: Other; p = 0.9146, t-test, 2 sided; Geometric Mean Ratio = 92.2, 90% CI 2-sided [23.0 to 368.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 160 mg Selpercatinib: Normal Hepatic Function vs 160 mg Selpercatinib: Severe Hepatic Impairment; Test type: Other; p = 0.7478, t-test, 2 sided; Geometric Mean Ratio = 119.6, 90% CI 2-sided [43.4 to 329.3] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: PK: Time to Reach Cmax (Tmax) of Selpercatinib
Description: PK: Tmax of Selpercatinib was reported.
Time Frame: as for outcome 1
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hour
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
hour | 2.00 [1.00 to 24.00] | 1.53 [1.00 to 2.03] | 2.00 [1.00 to 24.42] | 1.50 [1.00 to 3.00]

3. Primary Outcome: PK: Area Under the Concentration-time Curve (AUC), From Time 0 to the Last Observed Non-zero Concentration (AUC0-t) of Selpercatinib
Description: PK: AUC0-t was calculated using the linear trapezoidal rule for increasing and decreasing concentrations.
Time Frame: as for outcome 1
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/ mL)
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
hour*nanogram per milliliter (h*ng/ mL) | 17700 (65.0) | 20200 (43.1) | 14600 (74.0) | 27100 (33.7)
Statistical Analysis 1: Comparison: 160 mg Selpercatinib: Normal Hepatic Function vs 160 mg Selpercatinib: Mild Hepatic Impairment; Test type: Other; p = 0.4279, t-test, 2 sided; Geometric Mean Ratio = 126.1, 90% CI 2-sided [74.8 to 212.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 160 mg Selpercatinib: Normal Hepatic Function vs 160 mg Selpercatinib: Moderate Hepatic Impairment; Test type: Other; p = 0.8341, t-test, 2 sided; Geometric Mean Ratio = 92.4, 90% CI 2-sided [46.4 to 183.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 160 mg Selpercatinib: Normal Hepatic Function vs 160 mg Selpercatinib: Severe Hepatic Impairment; Test type: Other; p = 0.1159, t-test, 2 sided; Geometric Mean Ratio = 169.1, 90% CI 2-sided [97.1 to 294.6] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: PK: AUC Extrapolated to Infinity (AUC0-∞) of Selpercatinib
Description: PK: Area under the plasma concentration time curve extrapolated to infinity, calculated as AUC(0-t) + Ct/λZ, where Ct is the last measurable concentration and λZ is the apparent terminal elimination rate constant.
Time Frame: as for outcome 1
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/ mL)
Groups:
- Participants With Severe Hepatic Impairment: 160 mg Selpercatinib administered orally to participants with severe hepatic impairment per CP classification (CP Class C, score of 10 to 15) after at least a 2-hour fast on Day 1.
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
hour*nanogram per milliliter (h*ng/ mL) | 17700 (64.9) | 20200 (43.0) | 14700 (73.6) | 27300 (33.5)
Statistical Analysis 1: Comparison: 160 mg Selpercatinib: Normal Hepatic Function vs 160 mg Selpercatinib: Mild Hepatic Impairment; Test type: Other; p = 0.4289, t-test, 2 sided; Geometric Mean Ratio = 126.0, 90% CI 2-sided [74.8 to 212.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 160 mg Selpercatinib: Normal Hepatic Function vs 160 mg Selpercatinib: Moderate Hepatic Impairment; Test type: Other; p = 0.8322, t-test, 2 sided; Geometric Mean Ratio = 92.3, 90% CI 2-sided [46.5 to 183.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 160 mg Selpercatinib: Normal Hepatic Function vs Participants With Severe Hepatic Impairment; Test type: Other; p = 0.1131, t-test, 2 sided; Geometric Mean Ratio = 169.6, 90% CI 2-sided [97.6 to 294.6] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: PK: Percentage Extrapolation for AUC (%AUCextrap) of Selpercatinib
Description: PK: %AUCextrap of Selpercatinib was reported.
Time Frame: as for outcome 1
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: percentage of (%) of AUCextrap
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
percentage of (%) of AUCextrap | 0.422 (0.190) | 0.310 (0.197) | 0.373 (0.328) | 0.685 (0.379)

6. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (λz) of Selpercatinib
Description: PK: Apparent terminal elimination rate constant, where λZ is the magnitude of the slope of the linear regression of the log concentration versus-time profile during the terminal phase.
Time Frame: as for outcome 1
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour (1/h)
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
1/hour (1/h) | 0.0220 (61.4) | 0.0266 (39.8) | 0.0320 (29.0) | 0.0175 (28.8)

7. Primary Outcome: PK: Apparent Terminal Elimination Half-life (t1/2) of Selpercatinib
Description: PK: Apparent terminal elimination half-life (whenever possible), where t1/2 = natural log (ln)(2)/λZ.
Time Frame: as for outcome 1
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: hour
Groups:
- 160 mg Selpercatinib: Normal Hepatic Function: 160 mg selpercatinib administered orally to healthy participant after at least a 2-hour fast on Day 1.
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
hour | 36.4 (19.9) | 27.9 (12.2) | 22.4 (6.30) | 41.3 (13.5)

8. Primary Outcome: PK: Apparent Systemic Clearance (CL/F) of Selpercatinib
Description: CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided AUC (0-inf), expressed in liter/hour (L/hr).
Time Frame: as for outcome 1
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour (L/h)
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
Liters per Hour (L/h) | 9.03 (64.9) | 7.90 (43.0) | 10.9 (73.6) | 5.87 (33.5)

9. Primary Outcome: PK: Apparent Volume of Distribution During the Terminal Phase (Vd/F) of Selpercatinib
Description: PK: Vd/F was calculated as CL/F/λZ.
Time Frame: as for outcome 1
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
Liter (L) | 411 (51.5) | 297 (58.0) | 340 (68.6) | 336 (51.8)

10. Primary Outcome: PK: Mean Residence Time (MRT) of Selpercatinib
Description: PK: MRT represents the average time the drug (selpercatinib) stays in the body.
Time Frame: as for outcome 1
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
hour | 25.5 (21.9) | 23.3 (28.9) | 24.2 (39.2) | 34.3 (20.2)

11. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: Data presented are the number of participants who experienced SAEs considered by the investigator to be related to study drug administration. A summary of SAEs and all other non-serious Adverse Event(s) (AEs), regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Baseline up to Week 7
Population: All randomized participants who received at least one dose of study drug and had at least one post dose safety assessment.
Measure: Number; unit: participants
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 7
Description: All randomized participants who received at least one dose of study drug and had at least one post dose safety assessment.
Arm/Group | 160 mg Selpercatinib: Normal Hepatic Function | 160 mg Selpercatinib: Mild Hepatic Impairment | 160 mg Selpercatinib: Moderate Hepatic Impairment | 160 mg Selpercatinib: Severe Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/12 | 5/8 | 0/8 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 160 mg Selpercatinib: Normal Hepatic Function (N=12) | 160 mg Selpercatinib: Mild Hepatic Impairment (N=8) | 160 mg Selpercatinib: Moderate Hepatic Impairment (N=8) | 160 mg Selpercatinib: Severe Hepatic Impairment (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT05436912/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT05436912/SAP_001.pdf